CLINICAL TRIAL: NCT01933048
Title: Self-Administered Nasal Influenza Vaccine: Immunogenicity and Feasibility of Group Administration
Brief Title: Self-Administered Nasal Influenza Feasibility Study
Acronym: SNIF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IDCRP-070
Record Dates: First submitted 2013-08-08; First posted 2013-08-30 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Influenza
Keywords: influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthcare Worker Administration (Other): FluMist administered by a Healthcare Worker
  Interventions: Drug: FluMist
- Self-Administration (Experimental): FluMist self-administered by subject
  Interventions: Drug: FluMist

INTERVENTIONS:
Drug: FluMist — FluMist Intranasal Vaccine
  Other Names: influenza virus vaccine LAIV4

SUMMARY:
The purpose of this prospective, open-label clinical trial is to evaluate the immunogenicity of self-administered (SA) live, attenuated influenza vaccine (LAIV) in comparison with healthcare worker administered (HCWA) LAIV and to evaluate the feasibility of group self-administration of LAIV.

DETAILED DESCRIPTION:
This Phase IV, open-label, prospective clinical trial assesses SA-LAIV, testing whether the immunogenicity of SA-LAIV is non-inferior to that of HCWA-LAIV, as well as evaluating the feasibility of utilizing group administration for SA-LAIV. Subjects will be enrolled into one of two major treatment arms: HCWA-LAIV (Estimated N = 550) and SA-LAIV (Estimated N = 550). Enrollment into each major treatment arm will be stratified by study site. Enrollment in the HCWA-LAIV and SA-LAIV treatment arms may occur concurrently at each site. Subjects enrolling in the study will be randomized to HCWA or SA, and within the SA arm to either individual self-administration, or group administration. Specifically, following self-administration of LAIV to 190 individual subjects, 180 subjects will be vaccinated in 36 groups of 5 and 180 subjects will be vaccinated in 18 groups of 10. All vaccinations in the SA-LAIV arm will be given under the direction and supervision of a research staff member who is trained to administer LAIV vaccines. Following immunization all subjects will return for one visit at approximately 28 (± 7) days for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy, non-pregnant females
* 18-49 years of age
* Department of Defense beneficiary including active duty members
* Able to speak and understand English, and provide written informed consent

Exclusion Criteria:

* Known hypersensitivity to eggs, egg-proteins, gentamicin, gelatin, or arginine or life-threatening reactions to previous influenza vaccination
* Prior receipt of the 2012-2013 seasonal influenza vaccine for 2012-2013 season or prior receipt of the 2013-2014 seasonal influenza vaccine for 2013-2014 season
* Known clinical diagnosis of reactive airway disease, wheezing, or asthma (excluding exercise-induced asthma)
* Reported febrile upper respiratory illness (oral or tympanic temperature greater than 100°F or a subjective fever) at the time of or within the 24 hours prior to immunization
* Known to be pregnant, possibly pregnant or breast-feeding
* Known diagnosis of human immunodeficiency virus (HIV) infection, chronic active hepatitis B infection, or chronic hepatitis C infection
* History of Guillain-Barre Syndrome
* Household member known to be immunocompromised (either a known disease or disorder such as HIV, or other acquired or congenital immunodeficiency disorder, or taking systemic steroids (any dose) or high daily dose inhaled steroids, tumor necrosis factor-alpha inhibitors, or monoclonal antibodies used to treat autoimmune disease)
* Receipt of medications with activity against influenza A and/or B (ex: Tamiflu®, Relenza®, amantadine, or rimantadine) within 48 hours prior to vaccine administration
* Use of any oral or intravenous systemic steroids (any dose) or any daily dose inhaled steroids
* At the time of enrollment, any person who is trained to administer intranasal vaccines or who has been involved in any recurring role associated with the administration of intranasal vaccines to others in the clinic or military treatment facility (MTF)
* Prior participation in this research study
* Any acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, interfere with the evaluation of responses, or render the subject unable to meet the requirements of the protocol. These conditions may include, but are not limited to: history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); poorly controlled diabetes mellitus or patients with diabetes mellitus on insulin (subjects with well-controlled diabetes mellitus on oral agents may enroll as long there has been no dosage increase within the past 6 months); cardiac insufficiency, if heart failure is present; an arteriosclerotic event during the 6 months prior to enrollment (e.g., history of myocardial infarction, stroke, recanalization of femoral arteries, or transient ischemic attack).
* If the individual received a live virus vaccine (e.g., Varicella, Measles-Mumps-Rubella, Yellow Fever, Smallpox) in the past 4 weeks, they should wait 28 days before receiving LAIV. There is no reason to defer vaccination if the individual was vaccinated with an inactivated vaccine or if they have recently received blood or other antibody-containing blood products.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1077 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Burgess, MD, MPH, Study Director — Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - San Antonio Military Health System, Fort Sam Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Sharing of individual participant data (IPD) would require revisions and additional regulatory approval, that will not be pursued.

REFERENCES:
- [Derived] Burgess TH, Murray CK, Bavaro MF, Landrum ML, O'Bryan TA, Rosas JG, Cammarata SM, Martin NJ, Ewing D, Raviprakash K, Mor D, Zell ER, Wilkins KJ, Millar EV. Self-administration of intranasal influenza vaccine: Immunogenicity and volunteer acceptance. Vaccine. 2015 Jul 31;33(32):3894-9. doi: 10.1016/j.vaccine.2015.06.061. Epub 2015 Jun 25. PMID 26117150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment was conducted in San Antonio, Texas and San Diego, California.
Groups:
- Healthcare Worker Administration (HCWA): FluMist administered by a Healthcare Worker
- Self-Administration (SA): FluMist self-administered by subject
Period: Overall Study
Arm/Group | Healthcare Worker Administration (HCWA) | Self-Administration (SA)
Started | 548 | 529
Completed | 523 | 501
Not Completed | 25 | 28
Not completed — Lost to Follow-up | 15 | 18
Not completed — personal reasons | 1 | 1
Not completed — Protocol Violation | 7 | 8
Not completed — Physician Decision | 1 | 0
Not completed — unknown reasons | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthcare Worker Administration | Self-Administration | Total
Number analyzed (Participants) | 523 | 501 | 1024
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [26 to 38] | 28 [24 to 36] | 29 [25 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 141 | 298
  Male | 366 | 360 | 726
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 103 | 101 | 204
  Not Hispanic or Latino | 420 | 400 | 820
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 88 | 55 | 143
  White | 332 | 347 | 679
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 103 | 99 | 202
Region of Enrollment [Number; unit: participants]
  United States | 523 | 501 | 1024

OUTCOME MEASURES:

1. Primary Outcome: Post-vaccination Geometric Mean Titer (GMT) Ratios Between HCWA and SA Subjects
Time Frame: 28+/- 7 days post-vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titer ratio
Arm/Group | Healthcare Worker Administration | Self-Administration
Number analyzed (Participants) | 523 | 501
titer ratio
  A/H1N1 | 45.8 [41.1 to 51.1] | 48.7 [43.6 to 54.5]
  A/H3N2 | 45.5 [40.8 to 50.6] | 46.4 [41.6 to 51.8]
  B/Yamagata | 17.2 [15.9 to 18.6] | 17.8 [16.5 to 19.2]
  B/Brisbane (2013-2014 only; HCWA n=346; SA n=359) | 16.2 [14.7 to 17.9] | 14.7 [13.3 to 16.2]
Statistical Analysis 1: Comparison: Healthcare Worker Administration vs Self-Administration; A/H1N1; Test type: Non-Inferiority or Equivalence — non-inferiority; p = 0.43, Farrington-Manning Method; based on margin of 0.05
Statistical Analysis 2: Comparison: Healthcare Worker Administration vs Self-Administration; A/H3N2; Test type: Non-Inferiority or Equivalence — non-inferiority; p = 0.80, Farrington-Manning Method; based on margin of 0.05
Statistical Analysis 3: Comparison: Healthcare Worker Administration vs Self-Administration; B/Yamagata; Test type: Non-Inferiority or Equivalence — non-inferiority; p = 0.55, Farrington-Manning Method; based on margin of 0.05
Statistical Analysis 4: Comparison: Healthcare Worker Administration vs Self-Administration; B/Brisbane; Test type: Non-Inferiority or Equivalence — non-inferiority; p = 0.16, Farrington-Manning Method; based on margin of 0.05

2. Secondary Outcome: Difference and Proportion in Seroresponse of Subjects
Time Frame: 28+/- 7 days post-vaccination
Measure: Number; unit: participants
Arm/Group | Healthcare Worker Administration | Self-Administration
Number analyzed (Participants) | 523 | 501
participants
  A/H1N1 | 340 | 344
  A/H3N2 | 335 | 336
  B/Yamagata | 141 | 137
  B/Brisbane (2013-2014 only; HCWA n=346; SA n=359) | 84 | 79

3. Secondary Outcome: Difference and Proportion in Seroconversion of Subjects
Time Frame: 28+/- 7 days post-vaccination
Measure: Number; unit: participants
Arm/Group | Healthcare Worker Administration | Self-Administration
Number analyzed (Participants) | 523 | 501
participants
  A/H1N1 | 15 | 5
  A/H3N2 | 8 | 7
  B/Yamagata | 2 | 3
  B/Brisbane (2013-2014 only; HCWA n=346; SA n=359) | 23 | 14

4. Other Pre Specified Outcome: Feasibility of Self-administration Prior to Vaccine Administration
Time Frame: 28+/- 7 days post-vaccination
Measure: Number; unit: participants
Groups:
- Healthcare Worker Administration (HCWA): FluMist administered by a Healthcare Worker
  FluMist: FluMist Intranasal Vaccine
  Health care worker-administered (HCWA; n=523)
- Self-Administration (SA): FluMist self-administered by subject
  FluMist: FluMist Intranasal Vaccine
  Self-administered (SA)/singleton (n=178), SA/groups of 5 (n=163), and SA/groups of 10 (n=160).
Arm/Group | Healthcare Worker Administration (HCWA) | Self-Administration (SA)
Number analyzed (Participants) | 523 | 501
participants
  HCWA preferred method | 71 | 65
  SA preferred method | 132 | 129
  No preference | 320 | 307

5. Other Pre Specified Outcome: Feasibility of Self-administration Following Vaccine Administration
Time Frame: 28+/- 7 days post-vaccination
Population: Numbers include participants randomized to the SA group only.
Measure: Number; unit: participants
Arm/Group | Self-Administration (SA)
Number analyzed (Participants) | 501
participants
  HCWA preferred method | 29
  SA preferred method | 319
  No preference | 153

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Healthcare Worker Administration: This group includes healthcare worker administration of FluMist to subjects.
- Self-Administration: This group includes subjects who self-administered FluMist.
Arm/Group | Healthcare Worker Administration | Self-Administration
Serious Adverse Events (participants affected / at risk) | 2/548 | 3/529
Other Adverse Events (participants affected / at risk) | 13/548 | 24/529
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthcare Worker Administration (N=548) | Self-Administration (N=529)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1) — Hospitalized 4 days for pulmonary embolism. Not related to procedure. Relatedness=not probable.
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Hospitalized 4 days for deep vein thrombosis. Not related to procedure. Relatedness=not probable.
Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hospitalized overnight for hematoma after lipoma excision. Not related to procedure. Relatedness=unrelated.
Cholecystectomy (Hepatobiliary disorders) | 0 (0) | 1 (1) — Not related to procedure. Relatedness=unrelated
Hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hospitalization; chest/abdominal wall herniation from previous injury. Not related to procedure. Relatedness=unrelated.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthcare Worker Administration (N=548) | Self-Administration (N=529)
Syncope (Surgical and medical procedures) | 0 (0) | 2 (2) — Related to blood draw. Relatedness=definitely.
Nasal and chest congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Sinusitus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Cough and sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Headache (General disorders) | 0 (0) | 3 (3)
Tiredness and weakness (General disorders) | 2 (2) | 3 (3)
Nausea and diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Subjects were not followed for clinical outcomes during the influenza season.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No